CLINICAL TRIAL: NCT04486326
Title: Crofelemer for Functional Diarrhea
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Lembo, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P-000464
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — crofelemer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- crofelemer (Experimental): 125mg bid
  Interventions: Drug: Crofelemer
- placebo (Placebo Comparator): bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crofelemer — Crofelemer
  Other Names: mytesi
  Arms: crofelemer
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
The primary objectives of this study are to evaluate the clinical response of patients with diarrhea to crofelemer relative to placebo and evaluate the overall safety and tolerability of crofelemer in the treatment of diarrhea.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a man or woman aged 18 to 65 years, inclusive, at Screening.
2. Patient has functional diarrhea defined by the Rome IV criteria as loose (mushy) or watery stools ≥25% and hard or lumpy stools <25% of bowel movements
3. Patient has had a colonoscopy performed:

   1. Within 10 years prior to Prescreening if patient is at least 50 years of age (alternatively, a flexible sigmoidoscopy, double contrast barium enema, or CT colonography within the past 5 years is acceptable [see recommendations of the American Cancer Society])
   2. Since the onset (if applicable) of any of the following alarm features for patients of any age (see Spiller and Thompson, 2010 - i.e. Patient has documented weight loss within the past 6 months; Patient has nocturnal symptoms; Patient has a familial history of colon cancer; or patient has blood mixed with their stool (excluding any blood from hemorrhoids).
4. Patient has an average daily stool consistency score (BSS) of ≥5.5 on days without the use of an anti-diarrheal and at least 3 days with a BSS score ≥5 on a 1 to 7 scale over the week prior to randomization.
5. Patient has completed the daily diary on at least 6 of the 7 days during the week prior to randomization AND at least 11 of the 14 days during the 2 weeks prior to randomization.
6. Patient has not used loperamide rescue medication more than 4 days during the screening period.
7. Patient is not planning to change his/her usual diet and lifestyle during the course of the study.
8. Patient is willing to be compliant with study procedures including completing the daily diary during the screening period and throughout the study.
9. Patient must sign an informed consent document before the initiation of any study-related procedures indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. Patient has a history of inflammatory or immune-mediated GI disorders including inflammatory bowel disease (ie, Crohn's disease, ulcerative colitis, microscopic colitis) and celiac disease.
2. Patient has a predominant symptom of abdominal pain.
3. Patient has a history of diverticulitis within 3 months prior to screening. Patients with a history of diverticulosis are candidates for the study.
4. Patient has a history of intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (eg, aortoiliac disease).
5. Patient has any of the following surgical history:

   1. Any abdominal surgery within the 3 months prior to screening; or
   2. Patient has a history of major gastric, hepatic, pancreatic, or intestinal surgery (appendectomy, cholecystectomy, hemorrhoidectomy, or polypectomy greater than 3 months are allowed). For the purposes of this study, laparoscopic surgeries without complication are considered minor and non-exclusionary, provided the condition for which the surgery was performed was not exclusionary.
6. Patient has an unstable renal, hepatic, metabolic, or hematologic condition.
7. Patient has a history of human immunodeficiency virus infection.
8. Patient has a history of DSM-IV-TR-defined substance dependency, excluding nicotine and caffeine, within 2 years prior to Prescreening.
9. Patient has a history of alcohol abuse as defined by DSM-IV-TR, binge drinking as defined by the National Institutes on Alcohol Abuse and Alcoholism, or any medical treatment for alcohol-related co-morbidities, within 5 years prior to Prescreening. Recovered alcoholics who have not consumed alcohol over the 5 years prior to Prescreening are candidates for the study.
10. Patient has current (within 14 days of randomization) or expected use of any narcotic or opioid containing agents, tramadol
11. Patient is unable to swallow solid, oral dosage forms whole with the aid of liquid (patients may not chew, divide, dissolve, or crush the study drug).
12. Patient has received an investigational drug or used an investigational medical device within 30 days prior to randomization.
13. Patient has a known pregnancy or is breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Bristol Stool Form Scale | week 8
  measures stool consistency by type from 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lembo, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No